CLINICAL TRIAL: NCT07256327
Title: The Effects of Chiropractic on Kids With Sensory Processing Challenges: a Pilot Observational Study
Brief Title: Sensory Processing Challenges: a Pilot Observational Study
Acronym: SPD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Life University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I-0036
Record Dates: First submitted 2025-11-20; First posted 2025-12-01 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Sensory Processing Disorder
Keywords: Sensory Processing Disorder; Pediatric chiropractic care; autonomic nervous system

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Group (Experimental): 15 sessions of pediatric chiropractic care
  Interventions: Other: Chiropractic Care

INTERVENTIONS:
Other: Chiropractic Care — 15 sessions of normal and customary, fee-for-service, pediatric chiropractic care.

SUMMARY:
The main aims of this pilot observational study are to investigate the feasibility of implementing our novel assessment battery in tandem with normal and customary chiropractic care in a practice-based setting using a pediatric population with parent-reported SPD.

DETAILED DESCRIPTION:
Twenty (20) children with probable or definite parent-reported SPD (i.e., Short Sensory Profile (SSP) total scores ≤154) will be enrolled. More specifically, our primary outcomes are 1) enrollment, 2) eligibility, 3) tolerability, 4) adherence, and 5) retention. Secondary aims involve assessing the potential effects of subluxation-based chiropractic care on electrocardiography (ECG)-derived heart rate variability (HRV), bilateral weight distribution (BWD), and parent-reported outcomes (PROs). Data from this study will inform our lab regarding the feasibility of a larger study powered to assess the effectiveness of pediatric chiropractic care on clinical outcomes in a pediatric population with SPD.

ELIGIBILITY:
Inclusion Criteria:

* 5-12 years of age.
* SSP total scores ≤154

Exclusion Criteria:

* A known heart condition, including pacemakers
* Chiropractic care within the past 30 days

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2027-01-15 (Estimated); Study Completion 2027-01-15 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Enrolled | 1 year
  Proportion of approached parent/child pairs enrolled within the recruitment period time. This assesses uptake.
Number of Participants Eligible | 1 year
  Proportion of enrolled parent/child pairs who are eligible. This assesses eligibility.
Number of Participants Completing Assessments | 1 year
  Proportion of parent/child pairs able to complete all baseline assessments as directed. This assesses tolerability.
Number of Participants Completing Required Treatments | 1 year
  Proportion of parent/child pairs attending 15 sessions of chiropractic care within 10 weeks. This assesses adherence.
Number of Participants Remaining Enrolled | 1 year
  Proportion of parent/child pairs attending the final assessment session. This assesses retention.

SECONDARY OUTCOMES:
Changes in Electrocardiography Derived Heart Rate Variability | 1 year
  Change from baseline heart rate variability (HRV) using the MindWare mobile system. The device acquires lead-I electrocardiography (ECG) to derive a single HRV metric (RMSSD) representing autonomic regulation.
Changes in Bilaterial Weight Distribution | 1 year
  Change from baseline bilateral weight distribution utilizing a Wii Fit Balance Board, which tracks the percentage of weight borne by each leg.
Changes in Short Sensory Profile (SSP) | 1 year
  Change from baseline SSP. The SSP is a 38-item parent-report designed to assess a child's responsiveness to sensory stimuli including tactile sensitivity, taste/smell sensitivity, and visual/auditory sensitivity.
Change in Pediatric Autonomic Symptom Scales (PASS) | 1 year
  Change from baseline PASS. The PASS is an 80-item parent-report questionnaire designed to assess autonomic function in children across four main subscales: 1) mood, behavior, and emotion; 2) secretomotor/sensory integration; 3) urinary/gastrointestinal systems; 4) circulation, thermoregulation, sleep, and breathing.

IPD SHARING:
Plan to Share IPD: No